CLINICAL TRIAL: NCT01214304
Title: Aromatherapy With Lavender Oil to Reduce Pain and Anxiety During Cervical Colposcopy: A Randomized, Controlled Trial
Brief Title: Aromatherapy to Reduce Pain and Anxiety During Cervical Colposcopy
Acronym: Lavender Colpo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Collaborators: American Academy of Family Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20100154H
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Colposcopy
Keywords: Colposcopy
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lavender Scent (Placebo Comparator): Patients will receive aromatherapy with a fake lavender scent (placebo) which will be initiated 5 minutes prior to the procedure and continued until the conclusion of the procedure.
  Interventions: Other: Lavender Scent
- Essential Lavender Oil (Experimental): Patients will receive essential Lavender Oil which will be initiated 5 minutes prior to the procedure and continued until the conclusion of the procedure.
  Interventions: Other: Essential Lavender Oil

INTERVENTIONS:
Other: Essential Lavender Oil — Aromatherapy with essential lavender oil will be initiated 5 minutes prior to the procedure and continued until the conclusion of the procedure (patient dressed and ready to leave the room). The essential lavender oil and will be administered by fan diffuser.
  Arms: Essential Lavender Oil
Other: Lavender Scent — Aromatherapy with a fake lavender scent (placebo) will be initiated 5 minutes prior to the procedure and continued until the conclusion of the procedure (patient dressed and ready to leave the room). The fake lavender scent will be administered by fan diffuser.
  Arms: Lavender Scent

SUMMARY:
The purpose of this study is to determine whether aromatherapy with lavender oil compared to placebo lowers anxiety levels in women during colposcopy.

DETAILED DESCRIPTION:
Aromatherapy is a modality that might reduce anxiety. Women experience high levels of anxiety and negative emotional responses at all stages of cervical cancer screening. High levels of anxiety before and during colposcopy can be bad. If lavender oil aromatherapy reduces anxiety, then simple use of this modality may improve experiences during colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* All women at least 18 yrs of age undergoing colposcopy who have not previously participated in this protocol.

Exclusion Criteria:

* age <18 years
* pregnancy
* breastfeeding
* asthma
* poor sense of smell
* allergy to one of the essential oils
* consumption of any analgesic
* short-term anxiolytic (i.e. benzodiazepines) or chronic anxiolytic medications (i.e. SSRI)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain Level | 8 months
  Patients will be measured on an 11 point scale from 0 to 10 on their pain Level.

SECONDARY OUTCOMES:
Anxiety Level | 8 months
  Patients will be measured on an 11 point scale from 0 to 10 on their anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, M.D., Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Las Vegas, Nevada, United States